CLINICAL TRIAL: NCT04485208
Title: Open Label Study for the Use of Focused Transcranial Ultrasound for Treatment of Neuropathic Pain
Brief Title: Focused Ultrasound for the Treatment of Neuropathic Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Neurological Associates of West Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: fUS_NeuropathicPain
Record Dates: First submitted 2020-07-21; First posted 2020-07-24 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Active (Experimental): Patients will undergo ten to thirty minutes of transcranial ultrasound treatment. The sonification device will be aimed at the thalamus. Targeting will include reference to scalp fiducials based on the obtained MRI; confirmation of target accuracy will either be obtained by Doppler waveform confirmation or optical tracking technology which co-registers patient neuroimaging with real space.
  Interventions: Device: Focused Ultrasound

INTERVENTIONS:
Device: Focused Ultrasound — The DWL Doppler ultrasound device enables visual and auditory waveform confirmation of the anterior cerebral artery, and optical tracking technology (e.g., AntNeuro Visor2™ system) may be used in tandem with the Brainsonix Pulsar 1002 ultrasound device to track a patient's brain in virtual space as well as their physical location, thereby ensuring accurate placement.

SUMMARY:
A possible treatment approach for neuropathic pain would employ a process designed to promote healthier function of the ventral posteromedial (VPM) and ventral posterolateral (VPL) thalamic nuclei. This study is designed to employ focused ultrasound technology to target the VPM and VPL thalamus among participants with ongoing neuropathic pain syndromes to evaluate for tolerability and early efficacy.

DETAILED DESCRIPTION:
The present open-label study is being undertaken to evaluate focused transcranial ultrasound therapy as an intervention for patients with neuropathic pain. The subjects in this research study will be recruited through medical practice. Participants who are enrolled will undergo 8 consecutive weekly ultrasound sessions. Targeting for treatment will be based on patient MRI scans using stereotaxic techniques.

ELIGIBILITY:
Inclusion Criteria:

* History of neuropathic pain (onset, location, intensity, duration, quality, aggravating factors)
* Confirmation of nervous system injury through imaging or negative or positive sensory signs confined to the corresponding bodily area
* Failure from at least 3 pharmacological treatments (e.g., antidepressants, anticonvulsants, opioids)
* At least 18 years of age

Exclusion Criteria:

* Subjects unable to give informed consent
* Subjects who would not be able to lay down without excessive movement in a calm environment
* Pregnancy, women who may become pregnant or are breastfeeding
* Subjects with scalp rash or open wounds on the scalp (for example from treatment of squamous cell cancer)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-06-30 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Brief Pain Inventory (BPI) | Baseline
  Self-report measure containing a composite pain score and functional interference score. The pain subscale contains 4 questions, each with answers ranging from 0 'no pain' to 10 'pain as bad as you can imagine.' Total possible score for the pain subscale is 40 points. The functional/interference subscale contains 7 questions, with each answer ranging from 0 'does not interfere' to 10 'completely interferes.' The maximum possible score for the interference subscale is 70 points. The total overall composite BPI score is out of 100 maximum points. A clinical improvement is considered a decrease in BPI overall composite score by at least 30% from baseline.
Numeric Pain Rating Scale (NPRS) | Baseline
  The NRPS is a unidimensional measure of pain intensity for adults. The 11-point numeric scale ranges from '0' representing 'no pain' to 10 representing 'worst possible pain.' The NPRS can be administered verbally or graphically for self-completion. The respondent is asked to indicate the numeric scale value that best describes the intensity of their pain within the last 24-hours. Clinical improvement is denoted by at least 3 points improvement.
Patient Health Questionnaire (PHQ-9) | Baseline
  The PHQ-9 is a 9-item, self-report questionnaire to evaluate for depressive symptoms. Each question asks the patient if they have experienced a particular depressive symptom over the past two weeks. Answers may range from "0" (not at all), "1" (several days/week), "2" (more than half of the days), and "3" (nearly every day). Maximum total score is 27 points. A higher score indicates more severe depressive symptoms. A reduction in total score by at least 30% is considered clinically meaningful.

SECONDARY OUTCOMES:
Brief Pain Inventory (BPI) | Post Final Treatment (8 weeks from baseline)
  Self-report measure containing a composite pain score and functional interference score. The pain subscale contains 4 questions, each with answers ranging from 0 'no pain' to 10 'pain as bad as you can imagine.' Total possible score for the pain subscale is 40 points. The functional/interference subscale contains 7 questions, with each answer ranging from 0 'does not interfere' to 10 'completely interferes.' The maximum possible score for the interference subscale is 70 points. The total overall composite BPI score is out of 100 maximum points. A clinical improvement is considered a decrease in BPI overall composite score by at least 30% from baseline.
Numeric Pain Rating Scale (NPRS) | Post Final Treatment (8 weeks from baseline)
  The NRPS is a unidimensional measure of pain intensity for adults. The 11-point numeric scale ranges from '0' representing 'no pain' to 10 representing 'worst possible pain.' The NPRS can be administered verbally or graphically for self-completion. The respondent is asked to indicate the numeric scale value that best describes the intensity of their pain within the last 24-hours. Clinical improvement is denoted by at least 3 points improvement.
Patient Health Questionnaire (PHQ-9) | Post Final Treatment (8 weeks from baseline)
  The PHQ-9 is a 9-item, self-report questionnaire to evaluate for depressive symptoms. Each question asks the patient if they have experienced a particular depressive symptom over the past two weeks. Answers may range from "0" (not at all), "1" (several days/week), "2" (more than half of the days), and "3" (nearly every day). Maximum total score is 27 points. A higher score indicates more severe depressive symptoms. A reduction in total score by at least 30% is considered clinically meaningful.

CONTACTS AND LOCATIONS:
Overall Officials: Sheldon Jordan, MD, Principal Investigator — Neurological Associates of West Los Angeles
Locations (1):
- Neurological Associates of West LA, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cohen SP, Mao J. Neuropathic pain: mechanisms and their clinical implications. BMJ. 2014 Feb 5;348:f7656. doi: 10.1136/bmj.f7656. PMID 24500412
- [Background] Jang SH, Kim J, Lee HD. Delayed-onset central poststroke pain due to degeneration of the spinothalamic tract following thalamic hemorrhage: A case report. Medicine (Baltimore). 2018 Dec;97(50):e13533. doi: 10.1097/MD.0000000000013533. PMID 30558012
- [Background] Klit H, Finnerup NB, Jensen TS. Central post-stroke pain: clinical characteristics, pathophysiology, and management. Lancet Neurol. 2009 Sep;8(9):857-68. doi: 10.1016/S1474-4422(09)70176-0. PMID 19679277
- [Background] Kramer PR, Strand J, Stinson C, Bellinger LL, Kinchington PR, Yee MB, Umorin M, Peng YB. Role for the Ventral Posterior Medial/Posterior Lateral Thalamus and Anterior Cingulate Cortex in Affective/Motivation Pain Induced by Varicella Zoster Virus. Front Integr Neurosci. 2017 Oct 16;11:27. doi: 10.3389/fnint.2017.00027. eCollection 2017. PMID 29089872
- [Background] Krause T, Brunecker P, Pittl S, Taskin B, Laubisch D, Winter B, Lentza ME, Malzahn U, Villringer K, Villringer A, Jungehulsing GJ. Thalamic sensory strokes with and without pain: differences in lesion patterns in the ventral posterior thalamus. J Neurol Neurosurg Psychiatry. 2012 Aug;83(8):776-84. doi: 10.1136/jnnp-2011-301936. Epub 2012 Jun 13. PMID 22696587
- [Background] Mauguiere F, Desmedt JE. Thalamic pain syndrome of Dejerine-Roussy. Differentiation of four subtypes assisted by somatosensory evoked potentials data. Arch Neurol. 1988 Dec;45(12):1312-20. doi: 10.1001/archneur.1988.00520360030007. PMID 3196191
- [Background] Plotkin JL, Goldberg JA. Thinking Outside the Box (and Arrow): Current Themes in Striatal Dysfunction in Movement Disorders. Neuroscientist. 2019 Aug;25(4):359-379. doi: 10.1177/1073858418807887. Epub 2018 Oct 31. PMID 30379121
- [Background] Vartiainen N, Perchet C, Magnin M, Creac'h C, Convers P, Nighoghossian N, Mauguiere F, Peyron R, Garcia-Larrea L. Thalamic pain: anatomical and physiological indices of prediction. Brain. 2016 Mar;139(Pt 3):708-22. doi: 10.1093/brain/awv389. Epub 2016 Feb 8. PMID 26912644